CLINICAL TRIAL: NCT05589363
Title: A Comparison of the Analgesic Effects of Rectus Sheath and Transversus Thoracis Plane Blocks (ABC Blocks) Versus Saline Injection for Median Sternotomy: a Prospective, Randomized Controlled Trial.
Brief Title: ABC Blocks for Cardiac Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Budgetary issues
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00104058
Record Dates: First submitted 2022-09-28; First posted 2022-10-21 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: Anesthesia; Heart surgery; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABC block with bupivacaine and liposomal bupivacaine (Active Comparator): The study solution used in the active arm will comprise 20 mL of liposomal bupivacaine (266 mg) admixed with 40 mL of 0.25% bupivacaine HCl. The solution will be administered as bilateral parasternal blocks (40 mL) and bilateral epigastric rectus sheath blocks (20 mL).
  Interventions: Drug: ABC block with bupivacaine/liposomal bupivacaine
- ABC block with saline (Sham Comparator): The study solution used in the active arm will comprise 60 mL of 0.9% saline. The solution will be administered as bilateral parasternal blocks (40 mL) and bilateral epigastric rectus sheath blocks (20 mL).
  Interventions: Drug: ABC block with saline

INTERVENTIONS:
Drug: ABC block with bupivacaine/liposomal bupivacaine — Patients will be randomized to receive an ABC block using bupivacaine/liposomal bupivacaine solution
  Arms: ABC block with bupivacaine and liposomal bupivacaine
Drug: ABC block with saline — Patients will be randomized to receive an ABC block using normal saline
  Arms: ABC block with saline

SUMMARY:
This randomized blinded trial aims to evaluate the effect of parasternal intercostal and rectus sheath blocks ("anterior blocks for cardiac surgery" or ABC blocks) on postoperative recovery in patients undergoing median sternotomy for cardiac surgery. Subjects will be randomized to receive either local anesthetic (liposomal bupivacaine plus bupivacaine 0.25%) or saline sham block.

DETAILED DESCRIPTION:
Subjects will be randomized on the morning of surgery to receive either "anterior blocks for cardiac surgery" or "ABC blocks" using 60 mL of local anesthetic mixture (20 mL of liposomal bupivacaine plus 40 mL of 0.25% bupivacaine) or a sham saline ABC block (60 mL). All subjects will receive standard of care anesthetic regimen for their cardiac surgery at the discretion of his/her attending anesthesiologist. 40 mL of the solution will be administered in the parasternal intercostal space, and 20 mL will be placed in the rectus sheath in the epigastric region.

For the parasternal blocks, a linear high frequency ultrasound probe will be placed parasagitally at the T2-3 level approximately 3cm lateral to the mid-sternum, and all relevant structures will be identified, including the pectoralis major muscle, internal intercostal muscle, ribs, pleura, and any vasculature, including the internal mammary artery and vein. Color Doppler will be used confirm the location of vasculature.

After skin local anesthetic infiltration, a 10 cm 21G insulated block needle (Sonoplex, Pajunk Medical Systems, Norcross, GA) will be inserted from the inferior aspect of the ultrasound probe in a caudal to cranial direction and aligned with the ultrasound scanning plane (in-plane approach). In this way, both the needle shaft and tip can be visualized as the needle approaches the plane between the pectus major and intercostal muscles. The needle will be redirected as needed. Once satisfactory position of the needle time is confirmed and after frequent negative aspiration, 10 mL of study solution will be slowly injected. This injection will be repeated at the T4-5 interspace. Spread of local anesthetic will be documented in the appropriate plane in real time. This procedure will be performed bilaterally.

For the rectus sheath blocks, a linear high frequency ultrasound probe will be placed in a transverse position in the midline, just inferior to the xiphoid process. The probe will be moved laterally to visualize the lateral edge of the rectus abdominis muscle. A 10 cm 21G insulated block needle will be inserted from the lateral aspect of the ultrasound probe in a lateral to medial direction until visualized deep to the muscle immediately adjacent to the posterior rectus sheath. After negative aspiration, 10 mL of study solution will be slowly injected into this plane. This procedure will then be repeated on the contralateral side

All nerve blocks will be performed by a trainee supervised by an anesthesiologist experienced in regional anesthesia. The anesthesiology team and in the OR will be blinded to group allocation.

Subjects will receive a general anesthetic consistent with standard of care for cardiac surgeries at the discretion of his/her attending anesthesiologist. At the conclusion of the case, subjects will be extubated and/or transported to the ICU intubated. The decision to extubate the subject in the OR will be made at the discretion of the attending anesthesiologist.

Evaluation of acute postoperative pain intensity using a 0-10 visual analog scale (VAS) and opioid consumption will be undertaken at the following time points:

* 24 hours postoperatively
* 48 hours postoperatively Review of the medical chart will be made post-operatively to gather other data, including total intraoperative oral morphine equivalent consumption, cumulative opioid consumption at 48 hours, time to tracheal extubation, ICU length of stay, hospital length of stay, and time to first session with physical therapy. Occurrences of any adverse events reported by the subject or medical team will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for elective cardiac surgery involving primary median sternotomy
* Age 18-85 years of age
* BMI 18-50 kg/m2

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 30%
* Preoperative, intraoperative, or immediate post-operative placement of intra-aortic balloon pump or deployment of extra-corporeal membrane oxygenation (ECMO)
* Inability to understand or speak English
* Allergy to amide local anesthetic
* Contraindication to peripheral nerve block (e.g. local infection, previous trauma to the block site)
* Chronic opioid consumption (daily oral morphine equivalent of >20 mg) in the past three months
* Severe pulmonary disease
* Neurological deficit or disorder
* Suspected or known addition to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past two years
* Uncontrolled anxiety, schizophrenia, or other severe psychiatric disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption from extubation to 24 hours post-extubation | Extubation to 24 hr post-extubation
  Morphine equivalents administered between extubation and 24 hours post-extubation

SECONDARY OUTCOMES:
Worst pain at rest at 2 hours post-extubation | 2 hours post-extubation
  Pain intensity as measured on Numeric Pain Rating Scale (NRS-11) at 2 hours post-extubation. The NRS-11 ranges from '0' (no pain) to '10' (worst pain imaginable).
Worst pain at rest at 6 hours post-extubation | 6 hours post-extubation
  Pain intensity as measured on Numeric Pain Rating Scale (NRS-11) at 6 hours post-extubation. The NRS-11 ranges from '0' (no pain) to '10' (worst pain imaginable).
Worst pain at rest at 24 hours post-extubation | 24 hours post-extubation
  Pain intensity as measured on Numeric Pain Rating Scale (NRS-11) at 24 hours post-extubation. The NRS-11 ranges from '0' (no pain) to '10' (worst pain imaginable).
Worst pain at rest at 48 hours post-extubation | 48 hours post-extubation
  Pain intensity as measured on Numeric Pain Rating Scale (NRS-11) at 48 hours post-extubation. The NRS-11 ranges from '0' (no pain) to '10' (worst pain imaginable).
Cumulative opioid consumption from extubation to 48 hours post-extubation | Extubation to 48 hr post-extubation
  Morphine equivalents administered between extubation and 48 hours post-extubation
Time from end of case to tracheal extubation | End of operative case until patient extubated, up to 24 hours
  Time from end of surgical case (as defined by nursing record) until tracheal extubation
ICU length of stay | Postoperative from admission to ICU to discharge to floor, approximately 3 days
  Duration of time spent in cardiothoracic ICU from admission to discharge
Time to first session of physical therapy (PT) | 0-48 hours after surgical procedure
  Time from ICU admission until first session of physical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Manning, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No